CLINICAL TRIAL: NCT04863872
Title: Comparing the Effectiveness of Two Approaches to Preventing Severe Hypoglycemia
Brief Title: Comparing the Effectiveness of Two Approaches to Preventing Severe Hypoglycemia in Patients With Type 2 Diabetes (PHT2)
Acronym: PHT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IHS-2019C3-17889
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Severe Hypoglycemia
Keywords: Hypoglycemia; Self-management; Diabetes Mellitus, Type 2; Patient Education
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial comparing the effectiveness of 2 approaches for preventing severe hypoglycemia among participants with type 2 diabetes who are at risk for severe hypoglycemia. Participants were randomly assigned to one of two interventions: 1) Proactive Care Management, consisting of outreach from Kaiser Permanente Washington (KPWA) nurses using standard KPWA clinical tools; 2) the same Proactive Care Management plus MyHC-T2D, a structured educational intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Care Management (Active Comparator): Participants will receive one telephone nurse outreach call with follow up by the nurse or their primary care provider as clinically indicated.
  Interventions: Other: Proactive Care Management
- Proactive Care Management + MyHC-T2D education program (Experimental): Participants will receive the same telephone nurse outreach call with follow up as clinically indicated as the comparator arm and will in in additional be enrolled in a structured education program designed to improve hypoglycemia awareness and reduce severe hypoglycemia. The structured program will include 2 online group education sessions, 2 nurse follow up calls and use of glucose and hypoglycemia diaries, delivered over approximately 3 months.
  Interventions: Other: Proactive Care Management; Behavioral: MyHC-T2D education program

INTERVENTIONS:
Other: Proactive Care Management — Participants will receive one telephone nurse outreach call with follow up by the nurse or their primary care provider as clinically indicated.
Behavioral: MyHC-T2D education program — Participants will be enrolled in a structured education program designed to improve hypoglycemia awareness and reduce severe hypoglycemia. The structured program will include 2 online group education sessions, 2 nurse follow up calls and use of glucose and hypoglycemia diaries, delivered over approximately 3 months.
  Arms: Proactive Care Management + MyHC-T2D education program

SUMMARY:
Severe hypoglycemia is the most feared complication of medications used to lower blood glucose levels in patients with diabetes. Severe hypoglycemia, defined as plasma glucose low enough to require assistance, has been linked to poor health-related quality of life, emotional and interpersonal challenges, car accidents, serious falls, cardiovascular events, dementia, and death. Older adults with type 2 diabetes are particularly vulnerable to the complications of severe hypoglycemia. Each year, approximately 11% of patients with type 2 diabetes self-report severe hypoglycemia episodes. An estimated 14% of emergency hospitalizations of older Americans for adverse drug events implicate insulin and 11% implicate oral hypoglycemic agents. One in four diabetes-related hospital admissions is for hypoglycemia.

This study will compare two ways to reduce severe hypoglycemia in people with type 2 diabetes. The two methods to be compared are:

1. Proactive care management. This will be a nurse outreach call which is similar to the usual care that people with type 2 diabetes get to reduce their risk of severe hypoglycemia, but given in advance rather than in response to a recent severe hypoglycemia event.
2. The same proactive care management (nurse outreach call) plus enrollment in MyHC-T2D, a health education program aimed at improving awareness of hypoglycemia and preventing severe hypoglycemia. This program has been shown to reduce severe hypoglycemia in people with type 1 diabetes but has not been tested in persons with type 2.

Our hypothesis is that proactive care management plus MyHC-T2D will be more effective than proactive care management alone at preventing self-reported severe hypoglycemia in adults with type 2 diabetes at high risk for severe hypoglycemia. The primary outcome will be measured using surveys at the beginning of the study and 14-months later.

DETAILED DESCRIPTION:
This study is a two-arm, individually-randomized, comparative effectiveness study of two evidence-based approaches to preventing severe hypoglycemia. We will identify participants using Electronic Health Record (EHR) data. They will be identified for potential recruitment if they are age 18 and older, diagnosed with type 2 diabetes, receiving primary care at Kaiser Permanente Washington and have a current prescription for insulin or identified using an EHR-based risk stratification tool as being at intermediate to high risk for a severe hypoglycemia event. Within this population, we will recruit participants who either have impaired awareness of hypoglycemia or self-report a severe hypoglycemia event in the prior 12 months. Participants must be members of Kaiser Permanente Washington and identified by the study.

Following randomization, we will compare patients who receive proactive care management from nurses to patients receiving proactive care management plus MyHC-T2D, a structured educational intervention that reduces the frequency of severe hypoglycemia in individuals with type 1 diabetes. In both groups, we will use proactive care management to assess and provide evidence-based care for impaired awareness of hypoglycemia and other potential contributors to severe hypoglycemia risk.

Our primary outcome is participant-reported severe hypoglycemia, to capture all events, including those not involving clinical care. We will also examine biochemical measures of hypoglycemia measured using continuous glucose monitoring (CGM), participant-reported hypoglycemia awareness, fear of hypoglycemia, and emergency department visits and hospitalizations for severe hypoglycemia. We will conduct a process evaluation to assess the fidelity of implementation and clarify the causal pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with type 2 diabetes
* Receiving primary care at Kaiser Permanente Washington (KPWA)
* Enrollment in KPWA at baseline and planning to stay with a KPWA health plan for the next 6 months
* Current prescription for insulin or at intermediate to high risk for severe hypoglycemia episode using the hypoglycemia risk stratification tool developed by Karter et. al.
* History of severe hypoglycemia in the prior 12 months or impaired awareness of hypoglycemia

Exclusion Criteria:

* Inability to give informed consent
* Unable to speak or read English
* Inability or unwillingness to attend online or telephone educational sessions, follow up calls, or to complete outcome assessments
* Prior diagnosis of dementia, severe psychiatric conditions with psychosis, severe cognitive impairment
* Currently living in a nursing home or under hospice care
* Current use at baseline of Continuous Glucose Monitor
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Ralston, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karter AJ, Warton EM, Lipska KJ, Ralston JD, Moffet HH, Jackson GG, Huang ES, Miller DR. Development and Validation of a Tool to Identify Patients With Type 2 Diabetes at High Risk of Hypoglycemia-Related Emergency Department or Hospital Use. JAMA Intern Med. 2017 Oct 1;177(10):1461-1470. doi: 10.1001/jamainternmed.2017.3844. PMID 28828479
- [Background] Gold AE, MacLeod KM, Frier BM. Frequency of severe hypoglycemia in patients with type I diabetes with impaired awareness of hypoglycemia. Diabetes Care. 1994 Jul;17(7):697-703. doi: 10.2337/diacare.17.7.697. PMID 7924780
- [Background] Fitzgerald JT, Davis WK, Connell CM, Hess GE, Funnell MM, Hiss RG. Development and validation of the Diabetes Care Profile. Eval Health Prof. 1996 Jun;19(2):208-30. doi: 10.1177/016327879601900205. PMID 10186911
- [Derived] Ralston JD, Anderson M, Ng J, Bashir A, Ehrlich K, Burns-Hunt D, Cotton M, Hansell L, Hsu C, Hunt H, Karter AJ, Levy SM, Ludman E, Madziwa L, Omura EM, Rogers K, Sevey B, Shaw JAM, Shortreed SM, Singh U, Speight J, Sweeny A, Tschernisch K, Sergei Tschernisch S, Yarborough L. Preventing severe hypoglycemia in adults with type 2 diabetes (PHT2): Design, delivery and evaluation framework for a randomized controlled trial. Contemp Clin Trials. 2024 Apr;139:107456. doi: 10.1016/j.cct.2024.107456. Epub 2024 Jan 20. PMID 38253252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled based on identification from the Electronic Medical Record followed by outreach and telephone screening from January 2022 to January 2023. The first participant was enrolled on January 26, 2022 and the last participant was enrolled in January 2023.
Period: Overall Study
Arm/Group | Proactive Care Management | Proactive Care Management + MyHC-T2D Education Program
Started | 129 | 130
Completed | 118 | 112
Not Completed | 11 | 18
Not completed — Withdrawal by Subject | 4 | 15
Not completed — Death | 5 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proactive Care Management | Proactive Care Management + MyHC-T2D Education Program | Total
Number analyzed (Participants) | 129 | 130 | 259
Age, Customized [Count of Participants; unit: Participants]
  Age, categorical: Age less than 75 years | 92 | 92 | 184
  Age, categorical: Age 75 years and older | 37 | 38 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 81 | 157
  Male | 53 | 49 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 124 | 122 | 246
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 13 | 7 | 20
  White | 99 | 102 | 201
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 2 | 6 | 8
Hypoglycemic risk score [Count of Participants; unit: Participants] — Hypoglycemic risk score (low, moderate or high) is determined by a hypoglycemia risk stratification tool categorizing 12 month risk of hypoglycemia related utilization in individuals with type 2 diabetes using structured data from the electronic health record. From Karter et al, see Citation field in the Protocol section References.
  Participants
    Low | 60 | 61 | 121
    Moderate | 60 | 61 | 121
    High | 9 | 8 | 17
Impaired awareness of hypoglycemia [Count of Participants; unit: Participants] — Self-report of awareness of hypoglycemia using a 7-point Likert scale in response to the following question: "On a scale of 1 to 7, where 1 is always know and 7 is never know, how often do you know when your low blood sugars are beginning? The scale is 1 always, 7 never, with 4 in the middle. You can use any number 1, 2, 3, 4, 5, 6, 7." Participants were considered to have impaired awareness of hypoglycemia if they had a score of 4 or more. Question adapted from Gold et. al., see Citation field in the Protocol section References.
  Participants
    No impaired awareness | 24 | 12 | 36
    Impaired awareness | 104 | 118 | 222
    Missing | 1 | 0 | 1
Self report of any severe hypoglycemia in past 12 months [Count of Participants; unit: Participants] — Participants responded to the following standardized survey questions: "In the last 12 months, have you had low blood sugar that resulted in passing out or needing help from someone else? (For example, you were unable to treat yourself, were unconscious or were given glucagon or intravenous glucose)?" [if yes] "How many times did this happen (in the last 12 months)?" Question adapted from Fitzgerald et. al., see Citation field in the Protocol section References.
  Participants
    Zero | 85 | 97 | 182
    One or more | 44 | 32 | 76
    Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Severe Hypoglycemia
Description: Any self-reported severe hypoglycemia in prior 12 months
Time Frame: 14 months
Population: Participants included who completed the 14-month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Care Management | Proactive Care Management + MyHC-T2D Education Program
Number analyzed (Participants) | 118 | 112
Participants
  Zero | 99 | 99
  One or more | 19 | 13
Statistical Analysis 1: Comparison: Proactive Care Management vs Proactive Care Management + MyHC-T2D Education Program; Test type: Other — Difference; p = 0.27, Poisson regression; Poisson regression with binary primary outcome, estimated using Generalized Estimating Equations (GEE) and robust variance estimation; Risk Ratio (RR) = 0.72, 95% CI 2-sided [0.39 to 1.30]

ADVERSE EVENTS:
Time Frame: Self-reported adverse events were collected over 14 months from the time of the baseline survey through 14-month follow up. If a participant experienced an adverse event after informed consent was completed but before the participant started to receive the study intervention, the event was recorded and reported, but was determined as not related to the study intervention.
Description: Adverse events were collected using self-report open-ended survey questions at 6-, 10- and 14-month follow-up, and an open-ended question "Did you experience any difficulties with the Continuous Glucose Monitor (CGM)" after CGM data collection at baseline and 14 months. Study staff also recorded any adverse events reported spontaneously during scheduling calls. There were no differences between the ClinicalTrials.gov definitions and those used for this study.
Arm/Group | Proactive Care Management | Proactive Care Management + MyHC-T2D Education Program
All-Cause Mortality (participants affected / at risk) | 5/129 | 2/130
Serious Adverse Events (participants affected / at risk) | 46/129 | 56/130
Other Adverse Events (participants affected / at risk) | 39/129 | 54/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proactive Care Management (N=129) | Proactive Care Management + MyHC-T2D Education Program (N=130)
Stroke (Vascular disorders) | 1 | 5
Hospitalization, Not Otherwise Specified (General disorders) | 2 | 3
Myocardial infarction (Cardiac disorders) | 3 | 1
Hospitalization for syncope (General disorders) | 2 | 2
Hospitalization for fall (Injury, poisoning and procedural complications) | 0 | 4
Knee replacement (Surgical and medical procedures) | 2 | 2
Hospitalization for sepsis (Infections and infestations) | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hospitalization for urinary tract infection (Renal and urinary disorders) | 2 | 1
Pacemaker surgery (Surgical and medical procedures) | 1 | 2
Transient ischemic attack (Vascular disorders) | 3 | 0
Hospitalization for congestive heart failure (Cardiac disorders) | 1 | 1
Severe hypoglycemia (Endocrine disorders) | 1 | 1
Hospitalization for swelling in extremities, water retention (General disorders) | 1 | 1
Pancreatitis (Hepatobiliary disorders) | 0 | 2
Hospitalization for flue (Infections and infestations) | 0 | 2
Hospitalization for confusion (Nervous system disorders) | 1 | 1
Hospitalization for kidney problems (Renal and urinary disorders) | 2 | 0
Heart surgery (Surgical and medical procedures) | 1 | 1
Prostate surgery (Surgical and medical procedures) | 2 | 0
Surgery, Not Otherwise Specified (Surgical and medical procedures) | 1 | 1
Hospitalization for atrial flutter (Cardiac disorders) | 0 | 1
Heart valve transplant (Cardiac disorders) | 1 | 0
Heart problems (Cardiac disorders) | 0 | 1
Hospitalization for low heart rate (Cardiac disorders) | 0 | 1
Chest pain (Cardiac disorders) | 1 | 0
Gastrointestinal issues (Gastrointestinal disorders) | 1 | 0
Hospitalization for exhaustion (General disorders) | 1 | 0
Placed in Skilled Nursing Facility, Not Otherwise Spec (General disorders) | 1 | 0
Methotrexate toxicity (General disorders) | 0 | 1
Liver disease (Hepatobiliary disorders) | 0 | 1
Hospitalized for viral infection (Infections and infestations) | 0 | 1
Hospitalized for COVID-19 (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Broken leg (Injury, poisoning and procedural complications) | 0 | 1
Broken back (Injury, poisoning and procedural complications) | 0 | 1
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hospitalization for cyst in chest (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Slurred speech, confusion (Nervous system disorders) | 1 | 0
Hospitalized for kidney failure (Renal and urinary disorders) | 0 | 1
Hospitalized for high potassium (Renal and urinary disorders) | 1 | 0
Hospitalized for upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Knee surgery (Surgical and medical procedures) | 0 | 1
Laparotomy surgery (Surgical and medical procedures) | 0 | 1
Gall bladder surgery (Surgical and medical procedures) | 1 | 0
Lung surgery (Surgical and medical procedures) | 1 | 0
Carpal tunnel surgery (Surgical and medical procedures) | 0 | 1
Sinus surgery (Surgical and medical procedures) | 0 | 1
Hip surgery (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1
Hernia surgery (Surgical and medical procedures) | 0 | 1
Chin surgery (Surgical and medical procedures) | 0 | 1
Breast cancer surgery (Surgical and medical procedures) | 1 | 0
Gastric sleeve surgery (Surgical and medical procedures) | 0 | 1
Hospitalized for blood clots (Vascular disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Proactive Care Management (N=129) | Proactive Care Management + MyHC-T2D Education Program (N=130)
COVID-19 (Infections and infestations) | 9 | 12
Fall (Injury, poisoning and procedural complications) | 8 | 7
Itching with Continuous glucose monitor (Skin and subcutaneous tissue disorders) | 5 | 10
Hypoglycemia (Endocrine disorders) | 5 | 8
Bleeding with Continuous glucose monitor (Skin and subcutaneous tissue disorders) | 2 | 10
Discomfort with Continuous Glucose Monitor (Skin and subcutaneous tissue disorders) | 5 | 5
Confusion (Nervous system disorders) | 5 | 2

LIMITATIONS AND CAVEATS:
Both study groups received an intervention. Comparison to a group receiving usual care may have found different results. The proportion of individuals reporting a severe hypoglycemic event in the 12 months prior to baseline limited the ability to detect a change in the outcome at 14 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT04863872/Prot_SAP_000.pdf